CLINICAL TRIAL: NCT04137250
Title: Arthroscopic ACL Reconstruction: Hamstring Versus Quadriceps Tendon Autograft
Brief Title: Arthroscopic ACL Reconstruction: Hamstring Versus Quadriceps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, FELIX VILCHEZ CAVAZOS, Professor of Orthopedics and Traumatology, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR16-00008
Record Dates: First submitted 2017-03-10; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Anterior Cruciate Ligament Injury; Anterior Cruciate Ligament Rupture
Keywords: ANTERIOR CRUCIATE LIGAMENT; INJURY; HAMSTRING; AUTOGRAFT; QUADRICEPS
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a double-blind clinical trial with specific population, prospective, reproducible, comparative and longitudinal.
  It is proposed to study 28 patients, being randomly divided into two groups. We include patients of age between 18 years and 45 years, who have an anterior cruciate ligament injury diagnosed clinically and by image (magnetic resonance) and patients with or without associated meniscal injury, without previous reconstruction surgery and with previous informed Consent.
  We exclude patients with multiligamentous injury and/or those who have diagnosis of moderate or severe ostearthritis, chronic degenerative diseases (diabetes mellitus, hypertension) and contralateral ACL injury.
  We eliminate patients that for own initiative, wants to stop participating and those who didn't complete all follow-up appointments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hamstring (Active Comparator): It is the group in which the hamstrings are surgically removed to be used as an autograft for the reconstruction of the anterior cruciate ligament. The intervention will consist of make an incision on the medial side of the proximal portion of the leg approximately 3 centimeters to dissect by planes until the tendons of the hamstrings are located, which will be removed surgically with specialized instruments and the wound will be closed, for later These tendons be used as an autograft for the reconstruction of the anterior cruciate ligament.
  Interventions: Procedure: Hamstring
- Quadriceps tendon (Experimental): It is the group in which a portion of the quadriceps tendon will be surgically removed for later use as an autograft for the reconstruction of the anterior cruciate ligament. The intervention consisted in making an incision in the anterior aspect of the distal portion of the thigh of approximately 3 centimeters to dissect by planes until locating the membranous portion of the quadriceps tendon, from which will be removed a portion of surgical way with specialized instruments and the Wound will be closed, for later this tendon to be used as an autograft for the reconstruction of the anterior cruciate ligament.
  Interventions: Procedure: Quadriceps tendon

INTERVENTIONS:
Procedure: Hamstring — The intervention will consist of make an incision on the medial side of the proximal portion of the leg approximately 3 centimeters to dissect by planes until the tendons of the hamstrings are located, which will be removed surgically with specialized instruments and the wound will be closed, for later These tendons be used as an autograft for the reconstruction of the anterior cruciate ligament
  Arms: Hamstring
Procedure: Quadriceps tendon — orThe intervention consisted in making an incision in the anterior aspect of the distal portion of the thigh of approximately 3 centimeters to dissect by planes until locating the membranous portion of the quadriceps tendon, from which will be removed a portion of surgical way with specialized instruments and the Wound will be closed, for later this tendon to be used as an autograft for the reconstruction of the anterior cruciate ligament.
  Arms: Quadriceps tendon

SUMMARY:
The use of hamstrings and quadriceps autografts as an alternative option for reconstruction of the anterior cruciate ligament has good clinical results: however, both techniques have not been compared among them, which is why this study is intended. The use of quadriceps tendon autograft in anterior cruciate ligament repair presents similar or better results compared to autograft of the hamstrings. The objective of the study is to compare the clinical effectiveness of anterior cruciate ligament reconstruction between the use of quadriceps tendon autograft versus hamstring autograft.

DETAILED DESCRIPTION:
Methods Institution Patients attending the Orthopedics and Traumatology consult of the Hospital Universitario "Dr. Jose Eleuterio Gonzalez" of the Universidad Autonoma de Nuevo Leon.

Study design This is a double-blind , prospective, reproducible, comparative and longitudinal clinical trial with specific population.

It is proposed to study 28 patients, being randomly divided into two groups. Inclusion criteria: patients of age between 18 years and 45 years, with anterior cruciate ligament (ACL) injury diagnosed clinically and by magnetic resonance image and with or without associated meniscal injury, without previous reconstruction surgery and with previous informed Consent.

Exclusion criteria: multiligamentous injury and/or diagnosis of moderate or severe ostearthritis, chronic degenerative diseases (diabetes mellitus, hypertension) and contralateral ACL injury.

Elimination criteria: own initiative to stop participating and those who didn't complete all follow-up appointments.

Procedure Before surgery Detailed Informed Consent is performed to the patient before inclusion to the protocol Tegner Lysholm Knee Scoring Scale (evaluates the functionality of the knee and classifies them in grades with respect to its functional capacity) IKDC (evaluates knee ligament injuries, based on symptoms, sports activities and knee function) KOOS (evaluates knee sports injuries in young and middle-aged patients) Knee Society Score (pain, range of motion and injured knee stability) Cincinnati Knee Ligament Rating System (CKRS, assesses knee instability in ACL sports injuries) SF-12 (assesses patient's life quality) VAS (a subjective assesment of pain). Surgery The investigators will proceed to perform the anterior cruciate ligament reconstruction, both by the same surgeon, who will use the same technique in both groups, with the autograft in which the patient will have been randomly assigned.

After surgery all patients will be discharged previous warning signs explanation and several appointments in 2 weeks, 1 month, 3, 6 and 12 months after the procedure, for later evaluation scales, mentioned previously Statistical analysis In the sample size calculation, 14 patients per group are included using a mean equivalence formula, with 95% confidence and a power of 80%, estimating an equivalence of more less 2.5 on the Lysholm scale.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 45 years
* Anterior cruciate ligament injury diagnosed clinically and by image (magnetic resonance)
* Patients with or without associated meniscal injury
* Patients without previous ACL reconstruction surgery
* Patients with previous informed Consent.

Exclusion Criteria:

* Patients with multiligamentous injury
* Patients who have diagnosis of moderate or severe ostearthritis
* Patients with chronic degenerative diseases (diabetes mellitus, hypertension)
* Patients with contralateral ACL injury.

Elimination criteria

* Patients that for own initiative, wants to stop participating
* Patients who didn't complete all follow-up appointments.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
Lysholm knee score | up to 12 months (Baseline and 12 months)
  Assessment tool for the results of ACL reconstruction even though it only measures activities of daily living. Higher scores indicate a better outcome with fewer symptoms or disability.

SECONDARY OUTCOMES:
IKDC subjective score | up to 12 months (Baseline and 12 months)
  International Knee Documentation Committee Subjective Knee Form (IKDC) assess patients with a variety of knee disorders including ligamentous and meniscal injuries as well as patellofemoral pain and osteoarthritis. 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
SF-12 physical domain | up to 12 months (Baseline and 12 months)
  The 12-item Short Form Survey (SF-12) is a general health questionnaire that was first published in 1995 as part of the Medical Outcomes Study (MOS).
  Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
SF-12 mental domain | up to 12 months (Baseline and 12 months)
  The 12-item Short Form Survey (SF-12) is a general health questionnaire that was first published in 1995 as part of the Medical Outcomes Study (MOS).
  Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Flexion (degrees) | up to 12 months (Baseline and 12 months)
  Range of motion in degrees
Extension (degrees) | up to 12 months (Baseline and 12 months)
  Range of motion in degrees
Thigh circumference (cm) | up to 12 months (Baseline and 12 months)
  Circumference (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Vilchez, PhD, Principal Investigator — UANL
Locations (1):
- Facultad de Medicina UANL, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Lynch TS, Parker RD, Patel RM, Andrish JT; MOON Group; Spindler KP, Amendola A, Brophy RH, Dunn WR, Flanigan DC, Huston LJ, Jones MH, Kaeding CC, Marx RG, Matava MJ, McCarty EC, Pedroza AD, Reinke EK, Wolf BR, Wright RW. The Impact of the Multicenter Orthopaedic Outcomes Network (MOON) Research on Anterior Cruciate Ligament Reconstruction and Orthopaedic Practice. J Am Acad Orthop Surg. 2015 Mar;23(3):154-63. doi: 10.5435/JAAOS-D-14-00005. Epub 2015 Feb 9. PMID 25667401
- [Background] Prodromos CC, Fu FH, Howell SM, Johnson DH, Lawhorn K. Controversies in soft-tissue anterior cruciate ligament reconstruction: grafts, bundles, tunnels, fixation, and harvest. J Am Acad Orthop Surg. 2008 Jul;16(7):376-84. doi: 10.5435/00124635-200807000-00003. PMID 18611995
- [Background] Noyes FR, Butler DL, Grood ES, Zernicke RF, Hefzy MS. Biomechanical analysis of human ligament grafts used in knee-ligament repairs and reconstructions. J Bone Joint Surg Am. 1984 Mar;66(3):344-52. PMID 6699049
- [Background] Woo SL, Hollis JM, Adams DJ, Lyon RM, Takai S. Tensile properties of the human femur-anterior cruciate ligament-tibia complex. The effects of specimen age and orientation. Am J Sports Med. 1991 May-Jun;19(3):217-25. doi: 10.1177/036354659101900303. PMID 1867330